CLINICAL TRIAL: NCT07366736
Title: Monocentric Randomised Controlled Trial Assessing Cryocompression Following Total Knee Replacement
Acronym: CryoTKR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique des Cèdres (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-A01217-42
Record Dates: First submitted 2025-09-19; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Total Knee Anthroplasty; Cryotherapy; Compression
MeSH Terms: interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icepacks (Active Comparator): Directly following the surgery, the patient will go to the 'wake-up' area and will stay in the hospital for the next 1 to 3 days, during which the patients will use the icepacks to reduce inflammation. The patients will use icepacks for 4 hours consecutively directly following surgery.
  Interventions: Device: Cryotherapy
- Cryocompression (Experimental): Directly following the surgery, the patient will go to the 'wake-up' area and will stay in the hospital for the next 1 to 3 days, during which the patients will use the cryocompression to reduce inflammation. The patients will use cryocompression for 4 hours consecutively directly following surgery.
  Interventions: Device: Game Ready

INTERVENTIONS:
Device: Cryotherapy — Directly following the surgery, the patient will go to the 'wake-up' area and will stay in the hospital for the next 1 to 3 days, during which the patients will use the icepacks to reduce inflammation. The patients will use icepacks for 4 hours consecutively directly following surgery.
  Arms: Icepacks
Device: Game Ready — Directly following the surgery, the patient will go to the 'wake-up' area and will stay in the hospital for the next 1 to 3 days, during which the patients will use the cryocompression to reduce inflammation. The patients will use cryocompression for 4 hours consecutively directly following surgery.
  Arms: Cryocompression

SUMMARY:
Immediately following surgery, icepacks are commonly used to decrease inflammation and reduce pain and have demonstrated to decrease post-operative opioid consumption. New cryocompression devices have been introduced as a non-invasive and non-pharmacological modality used to manage acute inflammation and pain, demonstrating benefits in the post- operative setting promoting vasoconstriction, reducing blood flow and inflammation. The addition of compression may further decrease inflammation and pain, revealed in studies on anterior cruciate ligament reconstruction, total hip replacement, and lumbar fusion.

Recently, an RCT was published by Marinova et al. that compared cryocompression to icepacks following TKR in terms of pain on VAS, range of motion (ROM), knee circumference, and opioid consumption, but only found significant differences in extension ROM at day 1 and at 2 weeks. Due to the small sample size of Marinova et al. and high rates of losses to follow-up due to COVID-19, there remains doubt on the efficacy of cryocompression for TKR. Furthermore, cryocompression require additional investment in terms of cost to acquire the devices, and in time to train the hospital staff, and the devices may not be available for every patient. Finally, the authors are unsure how cryocompression affects wound healing in the short- and long-term.

The hypothesis was that both cryocompression and regular icepacks would grant equivalent pain on numeric rating scale at 48 hours postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years
* scheduled for primary TKR
* BMI <40 kg/m2
* who signed the informed consent and are willing to comply with the protocol requirements based on the investigator's judgment
* affiliated with a social security scheme
* with an ability to answer questionnaires and to communicate freely in French.

Exclusion Criteria:

* underwent revision TKR
* underwent bilateral TKR
* who cannot comply with the protocol requirements based on the investigator's judgment
* that are pregnant or breastfeeding
* with protected status under articles L1121-6, LL121-8 and L1122-2 of the French Public Health Code

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2027-07-27 (Estimated); Study Completion 2027-07-27 (Estimated)

PRIMARY OUTCOMES:
To compare post-operative pain between the intervention and the control group | 48 hours postoperatively
  Pain measured on numeric rating scale (NRS) at 48 hours postoperatively. 0 means no pain and 10 means severe pain.

SECONDARY OUTCOMES:
To compare post-operative pain during the study | 1, 3, and 9 months
  Pain measured on numeric rating scale (NRS), preoperatively, and postoperatively at 1, 3, and 9 months. 0 means no pain and 10 means severe pain.
To compare the evolution of joint function | preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 months
  Function assessed using the short version of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 months. It comprises five pain items (0-20), two stiffness items (0-8), and seventeen physical function items (0-68), using a 0-4 Likert scale (None to Extreme). The total score ranges from 0 (best) to 96 (worst).
To compare the evolution of mobility | preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 months
  Range of motion, including knee flexion and extension, measured using a goniometer, preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 months
To compare the incidence of oedema | preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 month
  Ipsilateral knee circumference and comparing it to the contralateral side, preoperatively, and postoperatively at 48 hours and at 1, 3, and 9 months
To compare wound healing | preoperatively, postoperatively at 48 hours and at 1, and 3 months
  Qualitative assessment: preoperatively, postoperatively assessed at 48 hours and at 1, and 3 months
To compare blood loss | preoperatively, and postoperatively at 24 hours, and 1 week
  Blood hemoglobin levels, preoperatively, and postoperatively at 24 hours, and 1 week
To compare pain killer consumption | at 48 hours, and at 1, 3 and 9 months
  Number, type and dosage of pain killers consumed at 48 hours, and at 1, 3 and 9 months
To compare quality of sleep | preoperatively, at 48 hours, and at 1, 3 and 9 months
  Using Pittsburgh Sleep Quality Index (PSQI) preoperatively, at 48 hours, and at 1, 3 and 9 months. This score involves summing seven component scores, each ranging from 0 (no difficulty) to 3 (severe difficulty), to get a global score from 0 to 21, with higher scores indicating poorer sleep quality, and a score > 5 generally suggesting significant sleep problems.
To compare safety of postoperative procedures | at 48 hours, and at 1, 3 and 9 months
  Incidence and severity of all adverse events related to the procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique des Cèdres, Échirolles, France

IPD SHARING:
Plan to Share IPD: No